CLINICAL TRIAL: NCT01708954
Title: A Randomized Phase II Trial of Erlotinib, Cabozantinib, or Erlotinib Plus Cabozantinib as 2nd or 3rd Line Therapy in Patients With EGFR Wild-Type NSCLC
Brief Title: Erlotinib Hydrochloride and Cabozantinib-s-Malate Alone or in Combination as Second or Third Line Therapy in Treating Patients With Stage IV Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01938; NCI-2012-01938 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-E1512; CDR0000741879; E1512 (Other: ECOG-ACRIN Cancer Research Group); E1512 (Other: CTEP); U10CA180820 (NIH); U10CA021115 (NIH)
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Results first posted 2016-12-01 (Estimated); Last update posted 2025-11-28 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Lung Non-Small Cell Carcinoma; Stage IV Lung Non-Small Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cabozantinib; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A (erlotinib) (Experimental): Patients receive erlotinib PO daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Erlotinib Hydrochloride; Other: Laboratory Biomarker Analysis
- Arm B (cabozantinib) (Experimental): Patients receive cabozantinib PO daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib S-malate; Other: Laboratory Biomarker Analysis
- Arm C (erlotinib+cabozantinib) (Experimental): Patients receive erlotinib as patients in Arm A and cabozantinib as patients in Arm B. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib S-malate; Drug: Erlotinib Hydrochloride; Other: Laboratory Biomarker Analysis
- Arm Z (erlotinib+cabozantinib; step II) (Experimental): Patients achieving disease progression in Arm A or Arm B may receive erlotinib and cabozantinib as patients in Arm C. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib S-malate; Drug: Erlotinib Hydrochloride; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL 184; XL-184; XL184
  Arms: Arm B (cabozantinib); Arm C (erlotinib+cabozantinib); Arm Z (erlotinib+cabozantinib; step II)
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: CP 358; CP-358; Cp-358,774; CP358; OSI 774; OSI-774; OSI774; Tarceva
  Arms: Arm A (erlotinib); Arm C (erlotinib+cabozantinib); Arm Z (erlotinib+cabozantinib; step II)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized phase II trial studies how well giving erlotinib hydrochloride and cabozantinib-s-malate alone or in combination works as second or third line therapy in treating patient with stage IV non-small cell lung cancer. Erlotinib hydrochloride and cabozantinib-s-malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether giving erlotinib hydrochloride together with cabozantinib-s-malate is more effective than erlotinib hydrochloride or cabozantinib-s-malate alone in treating non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the progression-free survival (PFS) associated with patients treated with erlotinib (erlotinib hydrochloride) versus (vs) erlotinib plus cabozantinib (cabozantinib-s-malate).

II. To compare the PFS associated with patients treated with erlotinib vs cabozantinib.

SECONDARY OBJECTIVES:

I. To evaluate overall survival in the three treatment arms. II. To evaluate best objective response rate in the three treatment arms. III. To define the toxicity associated with each regimen. IV. To conduct correlative science studies that will help to select predictive biomarkers of response to therapy, including mesenchymal-epidermal transition (MET) expression and potentially other tissue biomarkers, plasma biomarkers, and bone scans.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM A (erlotinib): Patients receive erlotinib orally (PO) daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B (cabozantinib): Patients receive cabozantinib PO daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM C (erlotinib+cabozantinib): Patients receive erlotinib as patients in Arm A and cabozantinib as patients in Arm B. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM Z: Patients achieving disease progression in Arm A or Arm B may receive erlotinib and cabozantinib as patients in Arm C. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Criteria:

* Tumor with a sensitizing mutation in epidermal growth factor receptor (EGFR), defined as follows:

  * EGFR mutation testing of tumor has been performed and did not demonstrate an EGFR tyrosine kinase inhibitor sensitizing mutation; at minimum, testing for EGFR exon 19 deletion and exon 21 L858R mutations must have been included; OR
  * EGFR mutation testing has been attempted and is inconclusive (for example, due to lack of sufficient deoxyribonucleic acid [DNA] yield); OR
  * EGFR mutation status is unknown but tumor is positive for at least one alternative driver mutation, i.e: Kirsten rat sarcoma viral oncogene homolog (KRAS) mutation, v-raf murine sarcoma viral oncogene homolog B (BRAF) mutation, human epidermal growth factor receptor 2 (HER2) mutation, ret proto-oncogene (RET) rearrangement/fusion, or one not listed following approval by the study chair prior to registration

Inclusion Criteria:

* INCLUSION CRITERIA STEP 1:
* Cytologically or histologically confirmed non-small cell lung carcinoma (NSCLC)
* Predominant non-squamous histology (patients with NSCLC not otherwise specified [NOS] are eligible); mixed tumors will be categorized by the predominant cell type; if small cell elements are present the patient is ineligible
* Stage IV disease (includes M1a, M1b, or recurrent disease), according to the 7th edition of the lung cancer TNM classification system
* Patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 criteria; baseline measurements and evaluation of all sites of disease must be obtained within 4 weeks prior to registration
* Prior to registration, the investigator/site must confirm that sufficient pathology material representative of patient's cancer is available for submission for MET immunohistochemical (IHC) testing
* Patients must have received one or two lines of prior chemotherapy (first line platinum-doublet based chemotherapy plus switch maintenance chemotherapy counts as one line of therapy); prior adjuvant chemotherapy for early stage disease does not count as one line of therapy if 12 months or greater elapsed between completion of adjuvant therapy and initiation of first-line systemic therapy; if less than 12 months elapsed, adjuvant chemotherapy counts as one line of therapy
* Any prior chemotherapy (based on administration schedule) must have been completed in greater than or equal to the time frames specified in the protocol
* Patients must have discontinued treatment with any other type of investigational agent >= 4 weeks prior to registration
* Patients must have recovered to baseline or Common Terminology Criteria for Adverse Events (CTCAE) v 4.0 =< grade 1 from toxicity due to all prior therapies except alopecia and other non-clinically significant adverse events (AEs)
* Patients with no known brain metastasis at baseline must have baseline brain imaging within 12 weeks prior to study registration not demonstrating brain metastases; patients with brain metastases at baseline must have baseline brain imagining within 4 weeks prior to study registration and meet all of the specific criteria for brain mets listed in the protocol
* Radiation related toxicities must have resolved to =< grade 1 prior to registration
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status between 0-2
* Patients must have an anticipated life expectancy greater than 3 months
* Acceptable bone marrow, renal and hepatic function within 2 weeks prior to registration as defined in the protocol
* Patients must have corrected QT interval calculated by the Fridericia formula (QTcF) =< 500 ms within 28 days before registration
* Patients must be able to swallow tablets
* INCLUSION CRITERIA STEP 2:
* Patients must have met all eligibility requirements for Step 1 at time of registration to Step 1 to be eligible for Step 2
* Patients must have radiographic progressive disease per RECIST v1.1 criteria after >= 2 courses of therapy on Arm A or Arm B
* Patients must be registered to Step 2 within 4 weeks of the last dose of treatment administration from Step 1
* Patients must have an ECOG performance status between 0-2
* Patients must have recovered to baseline (pre-Step 1) or CTCAE version 4.0 <= grade 1 from toxicity due to all prior therapies except alopecia and other non-clinically significant AEs

Exclusion Criteria:

* EXCLUSION CRITERIA STEP 1:
* Patients without sufficient pathology material representative of the patient's cancer (tumor block or 10 unstained slides)
* Prior erlotinib, other EGFR tyrosine kinase inhibitor therapy, vascular endothelial growth factor receptor (VEGFR) tyrosine kinase inhibitor therapy, Met tyrosine kinase inhibitor therapy, or Met monoclonal antibody (MetMAb); prior antibody therapy such as bevacizumab or cetuximab is allowed with a washout period depending on dosing interval and investigational nature
* Prior radiation therapy to the thoracic cavity, abdomen, or pelvis within 3 months prior to registration, to bone or brain metastasis within 14 days prior to registration, or to any other site within 28 days prior to registration
* History of the following: Clinically-significant gastrointestinal (GI) bleeding within 6 months prior to registration; Hemoptysis of >= 0.5 teaspoon (2.5 mL) of red blood within 3 months prior to registration; Any other signs indicative of pulmonary hemorrhage within 3 months prior to registration
* Radiographic or other evidence of the following within 28 days prior to registration: • Tumor invading the GI tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor; Cavitating pulmonary lesion(s); Tumor in contact with, invading or encasing any major blood vessels
* Psychiatric illness/social situations that would limit compliance with study requirements
* History of major thrombotic events (deep vein thrombosis [DVT] or pulmonary embolism [PE]) within 6 months prior to registration
* Concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, low molecular weight heparin (LMWH), thrombin or Factor Xa inhibitors, or antiplatelet agents (e.g., clopidogrel). (low dose aspirin [=< 81 mg/day] and prophylactic LMWH are permitted)
* Concomitant treatment of strong cytochrome P450 3A4 (CYP3A4) inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, and St. John's wort)
* Cardiovascular disorders including: Congestive heart failure (CHF): New York Heart Association (NYHA) class III (moderate) or class IV (severe) at the time of screening;
* Concurrent uncontrolled hypertension; Any history of congenital long QT syndrome; Any of the following within 6 months prior to registration:

  * Unstable angina pectoris
  * Clinically-significant cardiac arrhythmias
  * Stroke (including transient ischemic attack [TIA], or other ischemic event)
  * Myocardial infarction
* GI disorders particularly those associated with a high risk of perforation or fistula formation specified in the protocol
* Other disorders associated with a high risk of fistula formation including percutaneous endoscopic gastrostomy (PEG) tube placement within 3 months prior to registration
* Uncontrolled, significant, intercurrent or recent illness
* Prior malignancy within 2 years prior to registration which required systemic treatment or is currently active
* Pregnant or breast-feeding
* Patients with known human immunodeficiency virus (HIV) disease taking antiretroviral therapy
* Known chronic active hepatitis B
* EXCLUSION CRITERIA (STEP 2):
* Intervening anticancer treatment or major surgical procedure(s) between Step 1 and Step 2, except palliative radiation to the bone finishing >= 2 weeks prior to registration to Step 2
* Central nervous system (CNS) progression; patients with stable CNS disease are allowed
* Intercurrent illness or disease complication that the investigator believes would limit the ability to safely tolerate the combination of erlotinib and cabozantinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2013-02-13 (Actual); Primary Completion 2015-08-14 (Actual); Study Completion 2026-03-18 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joel W Neal, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (358):
- United States (358):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Memorial Medical Center, Modesto, California
  - Community Hospital of Monterey Peninsula, Monterey, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - IU Health Bloomington, Bloomington, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers-East, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - York Hospital, York Village, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Doylestown Hospital, Doylestown, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Einstein Medical Center Philadelphia, Philadelphia, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Texas Health Science Center at Tyler, Tyler, Texas
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - SSM Health Dean Medical Group - South Madison Campus, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

REFERENCES:
- [Derived] Neal JW, Dahlberg SE, Wakelee HA, Aisner SC, Bowden M, Huang Y, Carbone DP, Gerstner GJ, Lerner RE, Rubin JL, Owonikoko TK, Stella PJ, Steen PD, Khalid AA, Ramalingam SS; ECOG-ACRIN 1512 Investigators. Erlotinib, cabozantinib, or erlotinib plus cabozantinib as second-line or third-line treatment of patients with EGFR wild-type advanced non-small-cell lung cancer (ECOG-ACRIN 1512): a randomised, controlled, open-label, multicentre, phase 2 trial. Lancet Oncol. 2016 Dec;17(12):1661-1671. doi: 10.1016/S1470-2045(16)30561-7. Epub 2016 Nov 4. PMID 27825638

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on February 7, 2013 and closed to accrual on July 1, 2014 with final accrual of 125 patients. Among these, a total of 20 patients registered to Step 2.
Groups:
- Arm A (Erlotinib): Patients receive erlotinib 150mg PO daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm B (Cabozantinib): Patients receive cabozantinib 60mg PO daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm C (Erlotinib+Cabozantinib): Patients receive erlotinib 150mg PO daily and cabozantinib 40mg PO daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Step 1
Arm/Group | Arm A (Erlotinib) | Arm B (Cabozantinib) | Arm C (Erlotinib+Cabozantinib)
Started | 42 | 40 | 43
Started Protocol Therapy | 40 | 40 | 39
Eligible and Treated | 38 | 38 | 35
Patients With MET Status Data Available | 30 | 32 | 24
Completed | 0 (Treatment continued until progressive disease or unacceptable toxicity.) | 0 (Treatment continued until progressive disease or unacceptable toxicity.) | 0 (Treatment continued until progressive disease or unacceptable toxicity.)
Not Completed | 42 | 40 | 43
Not completed — Disease progression | 26 | 17 | 14
Not completed — Adverse Event | 3 | 11 | 13
Not completed — Death | 3 | 2 | 3
Not completed — Withdrawal by Subject | 2 | 5 | 3
Not completed — Other complicating disease | 0 | 2 | 0
Not completed — Crossed over to Step 2 | 2 | 0 | 0
Not completed — Symptomatic deterioration | 1 | 0 | 1
Not completed — Off-treatment reason not submitted | 1 | 1 | 1
Not completed — Ineligible or never received treatment | 4 | 2 | 8
Period: Step 2
Arm/Group | Arm A (Erlotinib) | Arm B (Cabozantinib) | Arm C (Erlotinib+Cabozantinib)
Started | 13 (Only patients with disease progression in Step 1 are eligible to register to Step 2.) | 7 (Only patients with disease progression in Step 1 are eligible to register to Step 2.) | 0 (Only patients with disease progression on Arms A and B were allowed to register to Step 2.)
Completed | 0 (Treatment continued until progressive disease or unacceptable toxicity.) | 0 (Treatment continued until progressive disease or unacceptable toxicity.) | 0
Not Completed | 13 | 7 | 0
Not completed — Disease progression | 9 | 4 | 0
Not completed — Adverse Event | 3 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Erlotinib) | Arm B (Cabozantinib) | Arm C (Erlotinib+Cabozantinib) | Total
Number analyzed (Participants) | 38 | 38 | 35 | 111
Age, Continuous [Median (Full Range); unit: years] | 68 [34 to 83] | 65 [46 to 88] | 63 [44 to 82] | 66 [34 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 17 | 61
  Male | 18 | 14 | 18 | 50

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from randomization to documented disease progression or death from any cause, whichever occurred first. Patients who had not experienced an event of interest by the time of analysis were censored at the date of last disease assessment.
Time Frame: Assessed every 3 months if patient is < 2 years from study entry; every 6 months if patient is 2 - 5 years from study entry, up to 5 years
Population: Eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Erlotinib) | Arm B (Cabozantinib) | Arm C (Erlotinib+Cabozantinib)
Number analyzed (Participants) | 38 | 38 | 35
months | 1.8 [1.7 to 2.2] | 4.3 [3.6 to 7.4] | 4.7 [2.4 to 7.4]
Statistical Analysis 1: Comparison: Arm A (Erlotinib) vs Arm C (Erlotinib+Cabozantinib); Test type: Superiority or Other; Hazard Ratio (HR) = 0.37, 80% CI 2-sided [0.25 to 0.53] — Hazard ratio of Arm C/Arm A
Statistical Analysis 2: Comparison: Arm A (Erlotinib) vs Arm B (Cabozantinib); Test type: Superiority or Other; Hazard Ratio (HR) = 0.39, 80% CI 2-sided [0.27 to 0.55] — Hazard ratio of Arm B/Arm A

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to death from any cause or date of last known alive.
Time Frame: as for outcome 1
Population: Eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Erlotinib) | Arm B (Cabozantinib) | Arm C (Erlotinib+Cabozantinib)
Number analyzed (Participants) | 38 | 38 | 35
months | 5.1 [3.3 to 9.3] | 9.2 [5.1 to 15.0] | 13.3 [7.6 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

3. Secondary Outcome: Proportion of Patients With Objective Response
Description: Objective response is defined as complete response (CR) or partial response (PR) evaluated using RECIST v 1.1. CR is defined as disappearance of all lesions and any pathological lymph nodes must have reduction in short axis to < 10 mm. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions and persistence of one or more non-target lesion(s).
Time Frame: as for outcome 1
Population: Eligible and treated patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Erlotinib) | Arm B (Cabozantinib) | Arm C (Erlotinib+Cabozantinib)
Number analyzed (Participants) | 38 | 38 | 35
proportion of participants | 0.03 [0.0009 to 0.141] | 0.11 [0.03 to 0.25] | 0.03 [0.001 to 0.15]

4. Secondary Outcome: Proportion of Patients With MET Positivity
Description: Submission of archival tissue for central MET IHC testing was required for this study, and total MET IHC testing was conducted at the Brigham and Women's Hospital using the c-Met clone CVD13 (arabbit polyclonal). Membranous and cytoplasmic staining were individually scored, and positivity was declared if MET was expressed in either the membrane or cytoplasm.
Time Frame: Assessed at baseline
Population: Eligible and treated patients who had sufficient samples for MET expression analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Erlotinib) | Arm B (Cabozantinib) | Arm C (Erlotinib+Cabozantinib)
Number analyzed (Participants) | 30 | 32 | 24
proportion of participants | 0.80 [0.61 to 0.92] | 0.81 [0.64 to 0.93] | 0.96 [0.79 to 0.999]

5. Secondary Outcome: Proportion of Patients With Worst Grade Toxicities of Grade 3 or Higher
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment
Population: All patients who received protocol therapy
Measure: Number (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm A (Erlotinib) | Arm B (Cabozantinib) | Arm C (Erlotinib+Cabozantinib)
Number analyzed (Participants) | 40 | 40 | 39
Proportion of participants | 0.325 [0.204 to 0.466] | 0.70 [0.560 to 0.817] | 0.718 [0.577 to 0.833]

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment
Groups:
- Arm Z (Erlotinib+Cabozantinib; Step 2): Patients achieving disease progression in Arm A or Arm B may receive erlotinib 150mg and cabozantinib 40mg as patients in Arm C. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm A (Erlotinib) | Arm B (Cabozantinib) | Arm C (Erlotinib+Cabozantinib) | Arm Z (Erlotinib+Cabozantinib; Step 2)
Serious Adverse Events (participants affected / at risk) | 13/40 | 28/40 | 28/39 | 12/20
Other Adverse Events (participants affected / at risk) | 35/40 | 40/40 | 38/39 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Erlotinib) (N=40) | Arm B (Cabozantinib) (N=40) | Arm C (Erlotinib+Cabozantinib) (N=39) | Arm Z (Erlotinib+Cabozantinib; Step 2) (N=20)
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 5 | 6 | 6 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 3 | 11 | 8
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 4 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 2 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 0
Lipase increased (Investigations) | 1 | 2 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0
Weight loss (Investigations) | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 1 | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 1 | 0 | 0
Dysphasia (Nervous system disorders) | 0 | 1 | 0 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 3 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 2 | 0 | 0
Vaginal fistula (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 10 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 3 | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Erlotinib) (N=40) | Arm B (Cabozantinib) (N=40) | Arm C (Erlotinib+Cabozantinib) (N=39) | Arm Z (Erlotinib+Cabozantinib; Step 2) (N=20)
Anemia (Blood and lymphatic system disorders) | 6 | 12 | 13 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 1 | 2 | 0 | 1
Edema limbs (General disorders) | 0 | 4 | 1 | 0
Fatigue (General disorders) | 20 | 27 | 32 | 13
Fever (General disorders) | 0 | 2 | 0 | 1
Pain (General disorders) | 0 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 9 | 10 | 3
Nail loss (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 6 | 6 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 2 | 7 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 23 | 6 | 25 | 9
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 4 | 6 | 3
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 4 | 3 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 5 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 10 | 2 | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 0 | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 4 | 4 | 3
Bloating (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 6 | 4 | 0
Diarrhea (Gastrointestinal disorders) | 24 | 23 | 31 | 15
Dry mouth (Gastrointestinal disorders) | 3 | 3 | 6 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 4 | 5 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 3 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 17 | 9 | 1
Nausea (Gastrointestinal disorders) | 8 | 19 | 17 | 4
Oral pain (Gastrointestinal disorders) | 0 | 2 | 4 | 1
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 4 | 5 | 11 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 2 | 0
Skin infection (Infections and infestations) | 1 | 2 | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 4 | 21 | 13 | 4
Alkaline phosphatase increased (Investigations) | 2 | 8 | 3 | 2
Aspartate aminotransferase increased (Investigations) | 8 | 26 | 17 | 10
Blood bilirubin increased (Investigations) | 5 | 5 | 4 | 2
Creatinine increased (Investigations) | 1 | 5 | 3 | 1
Lipase increased (Investigations) | 2 | 1 | 3 | 2
Lymphocyte count decreased (Investigations) | 1 | 5 | 5 | 2
Neutrophil count decreased (Investigations) | 0 | 2 | 2 | 0
Platelet count decreased (Investigations) | 1 | 14 | 8 | 2
Weight loss (Investigations) | 6 | 13 | 13 | 5
White blood cell decreased (Investigations) | 1 | 9 | 5 | 0
Anorexia (Metabolism and nutrition disorders) | 11 | 16 | 19 | 7
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 5 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 3 | 2 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 9 | 4 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 4 | 7 | 0
Hypokalemia (Metabolism and nutrition disorders) | 4 | 4 | 7 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 6 | 13 | 13 | 2
Hyponatremia (Metabolism and nutrition disorders) | 3 | 3 | 3 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 3 | 5 | 0
Dysgeusia (Nervous system disorders) | 6 | 12 | 11 | 6
Headache (Nervous system disorders) | 1 | 2 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 2 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 5 | 1 | 0
Conjunctivitis (Eye disorders) | 3 | 0 | 0 | 1
Dry eye (Eye disorders) | 2 | 2 | 2 | 0
Watering eyes (Eye disorders) | 1 | 1 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 6 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 2 | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 2 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 13 | 18 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 4 | 10 | 17 | 4
Thromboembolic event (Vascular disorders) | 2 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less